CLINICAL TRIAL: NCT01275326
Title: Indoor Air Quality and Infectious Aerosols in Health Care Facilities
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Hsing Chao, School of Public Health, Taipei Medical University
Other Study IDs: 99060
Record Dates: First submitted 2011-01-10; First posted 2011-01-12 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Indoor Air Quality; Infectious Aerosols
Keywords: Indoor Air Quality; Infectious Aerosols

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

SUMMARY:
Outbreaks of emerging and re-remerging infectious diseases are frequently reported internationally in recent years, mainly due to global climate change, close human-livestock contact in developing countries, and globalization. Thus prevention, monitoring and control of infectious diseases are in urgent need to protect public health. High exposure risk to various infectious agents in health care facilities is of special concern, especially to airborne and droplet-borne respiratory diseases. To protect the health of public and health care workers the investigators will conduct a study to monitor indoor air quality and essential infectious aerosols in hospital(s).

A questionnaire survey will be used to evaluate the relationships between employees' health and measured indoor environmental factors. The investigators will also examine whether the current indoor air quality recommendation of their country can reasonably reduce the risk of hospital infection. In addition, simple infectious aerosol indices will be established for future environmental management and monitoring in health care facilities.

ELIGIBILITY:
Inclusion Criteria:

* people who work in Health Care Facilities

Exclusion Criteria:

* none

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: people who work in Health Care Facilities
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2010-04; Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hsing Chao, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan